CLINICAL TRIAL: NCT00003752
Title: A Multicenter Phase II Evaluation of Targretin (Bexarotene) Capsules in Patients With Advanced Breast Cancer
Brief Title: Bexarotene in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: LIGAND-L1069-34; CDR0000066873 (Registry Identifier: PDQ (Physician Data Query)); MSKCC-99008; UMN-9808M00110
Record Dates: First submitted 1999-11-01; First posted 2004-05-25 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2007-05

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bexarotene

INTERVENTIONS:
Drug: bexarotene

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Randomized phase II trial to study the effectiveness of bexarotene in treating patients who have metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of oral bexarotene (LGD1069) at two different dose levels in patients with advanced breast cancer. II. Assess the safety and tolerability of this treatment regimen in this patient population. III. Evaluate the efficacy of oral bexarotene in terms of induction of differentiation and decreased aberrant cell proliferation in these patients.

OUTLINE: This is an open-label, randomized, multicenter study. Patients are stratified according to prior therapy for metastatic disease. Patients are randomized to one of two dose levels. All patients receive oral bexarotene once daily. Treatment continues in the absence of disease progression or unacceptable toxicity. Patients are followed every week for the first month, at weeks 6 and 8, then monthly thereafter.

PROJECTED ACCRUAL: A total of 84-180 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed metastatic breast cancer No CNS metastases No rapidly progressing visceral disease Previously irradiated lesions(s) may be designated as measurable indicator tumor(s) only if more than 6 months since radiotherapy, patient has no other measurable disease regrowth, and bidimensionally measurable regrowth is documented within 2 months prior to study Stratum 1 (hormonal): Must be hormone receptor positive (ER or PR) Prior hormonal therapy only allowed for metastatic disease Must have progressed on last hormonal regimen Must have at least one bidimensionally measurable tumor Stratum 2 (chemotherapy): Hormone receptor positive or negative Must have progressed on or after prior chemotherapy (1-2 regimens) for metastatic disease (bone marrow transplant counts as 2 regimens) Prior hormonal therapy allowed Must have at least one bidimensionally measurable tumor Stratum 3 (tamoxifen): Must be hormone receptor positive (ER or PR) and progressing on tamoxifen No symptomatic visceral metastasis if on adjuvant tamoxifen at time of systemic recurrence Must have at least one bidimensionally measurable tumor, or lytic bone lesion which measures at least one cm in diameter Hormone receptor status: See above

PATIENT CHARACTERISTICS: Age: Over 18 Menopausal status: Not specified Performance status: ECOG 0-2 OR Karnofsky 60-100% Life expectancy: At least 3 months Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Fasting triglycerides within normal range Hepatic: Bilirubin no greater than 1.5 times upper limit of normal (ULN) SGOT and/or SGPT no greater than 2.5 times ULN Concurrent medication with drugs that significantly alter hepatic metabolism (e.g., phenobarbital, phenytoin, oral azole antifungals) allowed only if dosage stable Renal: Creatinine less than 2 times ULN OR Creatinine clearance greater than 40 mL/min Concurrent medication with drugs that significantly alter renal metabolism (e.g., probenecid) allowed only if dosage stable Other: At least 5 years since any other prior invasive malignancy except basal cell and squamous cell carcinoma of the skin No serious concurrent illness that would prevent compliance No history of or clinically significant risk factors for developing pancreatitis Fasting triglycerides within normal range Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior monoclonal antibody HER2 therapy for metastatic disease allowed only if combined with chemotherapy or hormonal therapy and treatment failed No concurrent immunotherapy Chemotherapy: See Disease Characteristics At least 4 weeks since prior cytotoxic chemotherapy (at least 6 weeks since prior mitomycin or nitrosourea) No prior retinoid therapy for breast cancer At least 3 months since any other prior retinoid therapy except topical application for dermatological indications No concurrent chemotherapy Endocrine therapy: See Disease Characteristics At least 2 weeks since prior non-FDA approved hormonal therapy No other concurrent hormonal therapy except chronic low dose hormone replacement therapy or low dose corticosteroids for noncancer indication Radiotherapy: See Disease Characteristics Prior radiotherapy allowed Concurrent radiotherapy allowed only to non-indicator tumor(s) that do not represent new disease or disease progression Surgery: Prior surgery allowed Other: At least one month since prior investigational therapy (except hormonal) No other concurrent investigational therapy Concurrent medication with drugs that significantly alter hepatic metabolism (e.g., phenobarbital, phenytoin, oral azole antifungals) allowed only if dosage stable No more than 15,000 IU of vitamin A consumed daily

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 1998-10; Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George D. Demetri, MD, Study Chair — Dana-Farber Cancer Institute
Locations (30):
- United States (30):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Baptist Regional Cancer Institute - Jacksonville, Jacksonville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Louisiana State University School of Medicine, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Hematology Oncology Consultants Inc, Columbus, Ohio
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon-Minnie Pearl Cancer Center, Nashville, Tennessee
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Center, University of Virginia HSC, Charlottesville, Virginia

REFERENCES:
- [Result] Esteva FJ, Glaspy J, Baidas S, Laufman L, Hutchins L, Dickler M, Tripathy D, Cohen R, DeMichele A, Yocum RC, Osborne CK, Hayes DF, Hortobagyi GN, Winer E, Demetri GD. Multicenter phase II study of oral bexarotene for patients with metastatic breast cancer. J Clin Oncol. 2003 Mar 15;21(6):999-1006. doi: 10.1200/JCO.2003.05.068. PMID 12637463